CLINICAL TRIAL: NCT01913041
Title: An Epidemiology Survey on the Incidence of Perioperative Hypothermia of Patients Undergo Elective Operation With General Anaesthesia in Beijing Area
Brief Title: An Epidemiology Survey on the Incidence of Perioperative Hypothermia
Status: Completed | Type: Observational
Sponsor: Jie YI (Other)
Collaborators: 3M (Industry); Medical Consulting Center (Network)
Responsible Party: Sponsor-Investigator, Jie YI, Associate Professor, Peking Union Medical College Hospital
Organization: Peking Union Medical College Hospital (Other)
Other Study IDs: MDI0077
Record Dates: First submitted 2013-07-29; First posted 2013-07-31 (Estimated); Results first posted 2014-06-18 (Estimated); Last update posted 2014-07-16 (Estimated); Status verified 2014-07

CONDITIONS: Hypothermia
Keywords: perioperative hypothermia; Epidemiology; Tympanic temperature
MeSH Terms: conditions — Hypothermia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Investigation: This is an epidemiology study in which all the data from the subjects enrolled will be collected and analysis to investigate the current patient warming condition and actual perioperative hyperthermia rate in the elective operation with general anesthesia. During the whole procedure none intervention is administered.

SUMMARY:
* The purpose of this study is to understand and grasp the incidence rate of hypothermia during perioperative period of elective operations under general anaesthesia in Beijing.
* The purpose of this study is to carry out a subgroup analysis on the survey data and explore the high-risk factors for the incidence of hypothermia.

DETAILED DESCRIPTION:
This survey was anticipated to enroll 800 patients who underwent elective operations with general anaesthesia from 24 hospitals in Peking. After obtaining approval from the Ethical Committee related to research involving human subjects,the investigators will enroll the patients according to the inclusion and exclusion criterion. The tympanic temperature(measured by Braun PRO4000 Thermometer) will be monitored at the following time points respectively: arrived at waiting area, enter the OR room, 5 min before and after anesthesia induction, every 15 min during the operation, operation ended,arrived at PACU. Other information will also be collected, the investigators will record the type and dosage of anesthesia drug,duration of surgery and anesthesia, the patient warming method or if it is used.operation room temperature,the amount of the infusion of intravenous fluids and blood,etc. during the whole operation procedure. The other information will be followed up and recorded after the operation(within 30 days postoperation) which incudes ICU stays, hospital stays, incision infection, new cardiology events.etc.

The contract research organization will be delegated to do the site monitor once a week for each hospital participate the survey during the recruitment and perform the source data validation at the same time to review the related medical records,source data and the case report forms, etc.to ensure the data accuracy and completeness

Data management will be conduct through the whole survey procedure. EPIDATA3.1 software was used for compile the inputting procedure for data inputting and management. In order to guarantee the correctness of the data, two data managing staffs should input and verify the data independently.

SAS9.2 statistical analysis software was used for the calculation of all the statistical analyses. The number of cases, mean, standard deviation, median value, maximal value and minimal value should be calculated for the descriptions of the qualitative parameters. Number of cases and percentages are used for the descriptions on the classification parameters.Two side test is used for all the statistical tests, P<0.05 indicates that the difference is statistically significant (unless indicated otherwise), and 95% confidence is used as the confidence interval.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, no limitation on age
* Subject who will undergo elective surgery with general anaesthesia
* The duration of surgery is expected to be over 40 minutes
* The subject agreed to participate in the study and signed the informed

Exclusion Criteria:

* Central high fever caused by enter nerves system disease or condition, including that induced by cerebrovascular disease, cerebral trauma, cerebral surgeries, epilepsy and acute hydrocephalus
* Thermoregulation abnormalities including malignant hyperthermia (MHS) and neuroleptic malignant syndrome, hypothyroidism or hyperthyroidism diagnosed by substantial evidence
* Infectious fever
* Patients whose core temperature is higher than 38.5°C within 7 days before surgery
* Diseases or that may lead to inaccuracy in measurement, such as ear infection
* Surgeries with active cooling process during operation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who undergo elective surgery with general anaesthesia
Sampling Method: Probability Sample
Enrollment: 869 (Actual)
Dates: Start 2013-08; Primary Completion 2013-11 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yugung Huang, doctoral, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Dates of the recruitment period: From 2 Aug 2013 to 28 Nov 2013. Recruitment process: Random sample first and screening subjects according to the inclusion criteria and exclusion criteria, Assign ICF before enrollment.
Groups:
- Investigation Group: This is an epidemiology study in which all the data from the subjects enrolled will be collected and analysis to investigate the current patient warming condition and actual perioperative hyperthermia rate in the elective operation with general anesthesia. During the whole procedure none intervention is administered
Period: Overall Study
Arm/Group | Investigation Group
Started | 869
Completed | 830
Not Completed | 39
Not completed — Protocol Violation | 35
Not completed — Withdrawal by Subject | 3
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Population: 39 patients were eliminated for the reasons operation cancelled temporarily or volate the eligible criteria, so 830 participants for analysis was determined in the end.
Arm/Group | Investigation Group
Number analyzed (Participants) | 869
Age, Continuous [Median (Standard Deviation); unit: years] | 49.99 (16.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 347
  Male | 522
Region of Enrollment [Number; unit: participants]
  China | 869

OUTCOME MEASURES:

1. Primary Outcome: The Incidence of Perioperative Hypothermia
Description: Hypothermia incidence is defined as the percentage of the participants who occured hypothermia(Core temperature <36℃) accounts for the total amount of participants.
Time Frame: Perioperative period started from anesthesia induction to surgery ended
Population: Actually 869 patients are enrolled, among which 39 patients were eliminated for the reasons operation cancelled temporarily or violate the eligible criteria, so 830 participants for analysis was determined to be analyzed per protocol in the end.
Measure: Number; unit: Percentage of hypothermia participants
Arm/Group | Investigation Group
Number analyzed (Participants) | 830
Percentage of hypothermia participants | 39.8

ADVERSE EVENTS:
Groups:
- Observation Group: There is only one group, The main purpose of this investigation is to observe the hypothermia rate in elective operations under general anaesthesia in Peking in China.
Arm/Group | Observation Group
Serious Adverse Events (participants affected / at risk) | 0/869
Other Adverse Events (participants affected / at risk) | 0/869

LIMITATIONS AND CAVEATS:
In this study some information can hardly be completely collected such as wound infection incidence within 30 days postoperation, so further intervention study is needed to explore the relationship between hyperthermia and the potential complication.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days